CLINICAL TRIAL: NCT01135472
Title: Plasm Gastrin Concentrations in Response to Nexium Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08197
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: NEXIUM; HEALTHY VOLUNTEERS; BLOOD DRAW; to measure gastrin levels in healthy volunteers while taking nexium
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nexium (Experimental): ARM 1: NEXIUM 40MG ONCE DAILY, ARM 2: NEXIUM 40MG TWICE DAILY, ARM 3: NEXIUM 80MG TWICE DAILY
  Interventions: Drug: Esomeprazole Magnesium

INTERVENTIONS:
Drug: Esomeprazole Magnesium — NEXIUM 40MG ONCE DAILY FOR 7 DAYS WITH A 2 WEEK WASHOUT PERIOD, NEXIUM 40MG TWICE DAILY WITH A 2 WEEK WASHOUT PERIOD, NEXIUM 80MG TWICE DAILY WITH A 2 WEEK WASHOUT PERIOD.

SUMMARY:
This dose response study is proposed to explore the extent to which Nexium increases endogenous gastrin concentrations and to assess whether Nexium treatment may be useful in the setting of islet cell transplantation for type 1 diabetes to expand islet cells in vivo after transplant.

DETAILED DESCRIPTION:
Islet transplantation has been shown to effectively treat type 1 diabetes by stabilizing blood glucose control while reducing/eliminating the need for exogenous insulin injections. However, for reasons still not fully understood, islet graft function tends to decline with time after transplant. Gastrin has been identified as a growth factor capable of stimulating islet cell expansion. Proton pump inhibitors are known to increase endogenous gastrin concentrations. This dose response study is proposed to explore the extent to which Nexium increases endogenous gastrin concentrations in healthy volunteers and to assess whether Nexium treatment may be useful in expanding islet cells in patients with type 1 diabetes. Three Nexium dose levels will be tested to determine the optimal dose for increasing plasma gastrin levels. The effect of Nexium on plasma concentrations of glucose, insulin, c-peptide, glucagon, and somatostatin will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* healthy
* free of clinical signs of diabetes, peptic ulcer, liver or kidney disease,autoimmune disease, or any acute chronic infection.

Exclusion Criteria:

* history or clinical signs of diabetes
* history of liver or kidney disease
* positive H-pylori status
* currently using a proton pump inhibitor
* prior hypersensitivity to Nexium
* pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To measure the extent to which Nexium increases endogenous gastrin concentrations with 3 different treatment doses and least amount of side effects. | Every 3 days during treatment.
To measure the extent to which Nexium increases endogenous gastrin concentrations and returns to baseline levels during the two week non-treatment period. | Every 7 days during non-treatment period.

SECONDARY OUTCOMES:
To monitor the effect of Nexium on the plasma concentrations of glucose, insulin, c-peptide, glucagon, and somatostatin during 3 different treatment doses. | Every 3 days during treatment.
To monitor the effect of Nexium on the plasma concentrations of glucose, insulin, c-peptide, glucagon, and somatostatin during the two week non-treatment period. | Every 7 days during non-treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, Ph.D., Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States